CLINICAL TRIAL: NCT02595489
Title: A Pilot Study of Vitamin D in Boys With X-linked Adrenoleukodystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); ALD Connect, Inc. (Industry)
Responsible Party: Principal Investigator, Keith Van Haren, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23596; K23NS087151 (NIH)
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: Leukodystrophy; ABCD1; Demyelination; Inflammation; ALD; Vitamin D; Oxidative Stress; X- linked; Adrenoleukodystrophy
MeSH Terms: conditions — Adrenoleukodystrophy; Demyelinating Diseases; Inflammation | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: single-arm dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin D3 (Experimental): Single-arm, dose-escalation starting at 1,000 IU or 2,000 IU of vitamin D3 daily for a 6 month period, followed by a conditional titration up to 4,000 IU daily for at least 6 months thereafter. No placebo.
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Daily oral supplement provided by study investigators
  Other Names: vitamin D

SUMMARY:
In this pilot study, the investigators will assess the safety of two high-dose regimens of oral vitamin D supplementation and measure the effects of vitamin D supplementation on markers of oxidative stress and inflammation in the blood and brain of study participants before, during, and after taking vitamin D supplements.

The goal of the study is to establish research measures (i.e. biomarkers) and an optimal dose for vitamin D supplementation in boys with the X-linked adrenoleukodystrophy (ALD) genotype.

DETAILED DESCRIPTION:
Prior research suggests that higher vitamin D levels in the blood are associated with reduced brain inflammation among individuals with multiple sclerosis, a disease that is similar to the cerebral demyelinating form of ALD. However, serious side effects (e.g. hypercalcemia, kidney stones) can occur if vitamin D levels get too high.

The current study is designed to establish a safe dose of vitamin D for boys with ALD. Although the doses chosen for this study are expected to be safe, the investigators will monitor participants for early signs of vitamin D-related toxicity. The investigators will also examine whether or not vitamin D supplementation affects markers of oxidative stress and inflammation in the blood and brains of ALD boys.

The study requires participants to agree to at least one year of participation. Participants will be asked to take a vitamin D supplement every day, submit blood for analysis every 3 months in the first year, and visit their study center (Stanford University or the Kennedy Krieger Institute) every 6 months throughout the period of study.

Participants will be assigned a vitamin D dose based on bodyweight at entry. Starting doses will include 1,000 or 2,000 international units (IU) of vitamin D3 daily for a 6 month period, followed by a conditional increase to 2,000, 3,000, or 4,000 IU daily thereafter if vitamin D levels have not achieved a target threshold. The vitamin D supplements will be provided by the study. In keeping with the current standard of care for ALD boys aged 18mos - 25 years, participants will need to visit the study site every six months in order to complete a clinic visit and MRI of the brain with gadolinium. As part of this study, however, participants' will need to submit blood work every 3 months during the first year in order for the study investigators to ensure that the participants' calcium and vitamin D levels are in a safe range and to study the effects of vitamin D on markers in the blood. The MRI protocol during the first year will also include one additional sequence (magnetic resonance spectroscopy) in order to measure brain metabolites.

The data generated from this study are intended, in part, to help design a future, large-scale clinical trial to determine whether vitamin D supplementation is capable of reducing the risk of developing the cerebral demyelinating form of ALD.

ELIGIBILITY:
Criteria for enrollment to screening:

1. Molecular confirmation of X-linked ALD (VLCFA elevation & ABCD1 mutation) known in patient or immediate family member)
2. Male
3. Age 1.5yrs (i.e. 18mos) - 25yrs at screening

Criteria for assignment to drug:

1. Plasma 25-hydroxy vitamin D level ≤ 60ng/ml in past 30 days
2. MRI brain in past 6 months that is negative for evidence of active cerebral demyelination

Exclusion Criteria:

* history of liver or kidney disease
* history of nephrolithiasis
* history of hyperthyroidism
* history of ulcerative colitis, Crohn's disease, celiac disease
* taking medication interfering with gastrointestinal absorption
* contraindication or inability to complete MRI every 6 months

Ages: 18 Months to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Percent of patients with a plasma 25-OH vitamin D level in the target range (40-80ng/ml) at 12 months | Plasma 25-OH vitamin D will be measured at 12 months
  The investigators expect 100% of patients will be in the target range at 12 months (i.e. oral dose of 4000 IU daily)
Percent of patients with a plasma 25-OH vitamin D level in the target range (40-80ng/ml) at 6 months | Plasma 25-OH vitamin D will be measured at 6 months
  The investigators expect that 80% of patients will be in the target range 6 months (i.e. oral dose of 2000 IU daily)

SECONDARY OUTCOMES:
Correlation between appearance of gadolinium enhancing brain lesion on MRI and most recent plasma 25-OH vitamin D level | Brain MRI at baseline, 6, 12, 18, 24, 30, and 36 months study enrollment. Plasma 25-OH vitamin D levels at baseline, 3, 6, 9, 12, 18, 24, 30, 36 months of enrollment.
  For participants developing gadolinium enhancing lesions on MRI, the investigators will compare the most recent preceding 25-OH vitamin D level with the average 25-OH vitamin D level of participants in the study who did not develop gadolinium enhancing lesions. The investigators expect the development of gadolinium enhancing lesion on MRI will correlate with lower vitamin D levels. However, our current study is not sufficiently powered to measure this effect.
Change in protein carbonyl levels in whole blood at baseline and 12 months. | Measurements at baseline and 12months
  The investigators expect a decrease in whole blood protein carbonyl levels between baseline and 12 months.
Correlation between plasma 25-OH vitamin D and intracellular glutathione levels in peripheral monocytes | Measurements at baseline and 12 months
  The investigators will use flow cytometry to measure intracellular GSH in CD14+ monocytes from participants peripheral blood at baseline and 12 months. The investigators will measure plasma 25-OH vitamin at the same time points. The investigators expect a positive correlation between plasma vitamin D levels and monocyte GSH levels.
Change in glutathione (GSH) levels in blood | Measurements will be obtained at baseline, 6months, and 12months
  The investigators expect a positive correlation between plasma 25-OH vitamin levels and GSH levels in whole blood (measured by tandem mass spectroscopy).
Change in glutathione (GSH) levels in brain | Measurements will be obtained at baseline, 6months, and 12months
  The investigators will examine the correlation between 25-OH vitamin D levels in plasma and total GSH levels in occipital white matter (measured by single-voxel MR spectroscopy).
Occurrence of serious adverse events | Measurements will be obtained at baseline, 3months, 6months, 9months, 12months
  The investigators do not expect any participants to develop hypercalcemia (serum calcium >10.7mg/dl) or related serious adverse events (e.g. kidney stones) while taking 2000 IU or 4000 IU daily.
Change in plasma interleukin-8 levels | Measurements a baseline and 12 months
  The investigators expect a decrease in plasma IL-8 levels between baseline and 12 months
Change in plasma macrophage inflammatory protein-1b levels | Measurements at baseline and 12 months
  The investigators expect a decrease in plasma MIP-1b levels between baseline and 12 months
Change in plasma monocyte chemoattractant protein-1 levels | Measurements at baseline and 12 months
  The investigators expect a decrease in plasma MCP-1 levels between baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith Van Haren, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available to clinical investigators upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For up to 10 years following study completion
Access Criteria: Reasonable request via email to study PI (kpv@stanford.edu)

REFERENCES:
- See also: Stanford University Neurosciences Patient Registry for Clinical Trials — https://redcap.stanford.edu/surveys/?s=kCXDqU
- See also: Multiple Sclerosis and Neuroimmunology Clinical Trials — http://med.stanford.edu/neurology/divisions/neuroimmunology/clinicaltrials.html

DOCUMENTS (1):
  • Informed Consent Form (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT02595489/ICF_000.pdf